CLINICAL TRIAL: NCT05653076
Title: Hibiscus Sabdariffa Extract Effect on Neuromuscular Performance After Intense Resistance Exercise: a Randomized, Placebo-controlled, Crossover Study
Brief Title: Hibiscus Sabdariffa Extract Effect on Neuromuscular Performance
Acronym: RECUPERA-T
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Francisco Javier Osuna-Prieto, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1364-N-22
Record Dates: First submitted 2022-11-28; First posted 2022-12-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Neuromuscular Performance
Keywords: nutritional ergogenics; sport supplementation; anthocyanins; polyphenols; antioxidants; strength

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: triple-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Microcrystalline cellulose
  Interventions: Dietary Supplement: Hibiscus sabdariffa extract
- Hibiscus sabdariffa extract (Experimental): 520 mg of Hibiscus sabdariffa extract
  Interventions: Dietary Supplement: Hibiscus sabdariffa extract

INTERVENTIONS:
Dietary Supplement: Hibiscus sabdariffa extract — Daily supplementation with 520 mg of Hibiscus sabdariffa extract for 10 days.

SUMMARY:
Exercise-induced muscle damage (EIMD) is a transient problem that athletes face after performing more intense and/or prolonged exercise than they are used to. EIMD is accompanied by an increase in the production of reactive oxygen species and a decrease in the antioxidant capacity of the organism. This phenomenon decreases the performance capacity of athletes due to impaired muscle strength and range of motion. Among the strategies to reduce EIMD, the use of nutritional strategies rich in antioxidants such as polyphenols stands out. In this sense, the extract of Hibiscus sabdariffa is particularly rich in polyphenolic antioxidants, among which anthocyanins stand out. Previous studies have concluded that the administration of an extract of Hibiscus sabdariffa can prevent overtraining syndrome by reducing the levels of oxidizing agents and increasing the body's antioxidant defenses. However, despite the fact that Hibiscus sabdariffa extract has been shown to be safe for humans to ingest and have various health benefits, to our knowledge, no studies have evaluated its ability to minimize neuromuscular performance impairment that occurs after performing an intense session of strength training. Based on previous evidence, we hypothesize that supplementation with an extract of Hibiscus sabdariffa will improve neuromuscular performance after performing intense resistance exercise in young (18-35 years) and trained adults, with at least 1 year of experience training. strength. The design of this study is crossover, randomized and placebo controlled, where each individual will act as her own control. The neuromuscular performance parameters to be evaluated will be: i) explosive strength - main variable, in terms of countermovement jump height (CMJ); ii) the maximum dynamic force; and iii) the ability to change direction, all of them 24h and 72h after a high-intensity strength training session. If our hypothesis is confirmed, the results of our study would not only have an impact at a scientific level but also at a commercial level through the development of supplements and/or functional foods.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years.
* Body mass index: 18.5-30 kg/m2
* Be able to understand the instructions, objectives, and protocol of the study.
* Trained in some force sports discipline ≥1 year prior to the study and accustomed to carrying out the exercises of the evaluation protocol.

Exclusion Criteria:

* History of a major adverse cardiovascular event, renal failure, cirrhosis, eating disorder, polycystic ovarian syndrome, weight control surgery, type 2 diabetes mellitus, or HIV/AIDS.
* Any chronic pathology in which the intake of nutritional supplements is not recommended.
* Any condition that, in the investigator's judgment, impairs the ability to participate in the study or represents a personal risk to the participant.
* Use of medications that may affect the results of the study.
* Unstable body weight for 3 months prior to study start (>4 kg weight gain or loss)
* Routine use of teas/infusions/supplements rich in polyphenols.
* Pregnancy and lactation.
* Active tobacco or illicit drug use or history of treatment for alcohol abuse.
* To be on a special diet or prescribed for other reasons (eg celiac disease).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Explosive strength | 1 day (24h) after a bout of an intense resistance exercise
  It will be measured through the height of the countermovement jump (CMJ)
Maximal dynamic force | 1 day (24h) after a bout of an intense resistance exercise
  It will be measured by means of a CMJ with a load
Ability to change direction | 1 day (24h) after a bout of an intense resistance exercise
  It will be measured by means of a CMJ with a load

SECONDARY OUTCOMES:
Explosive strength | 3 days (72h) after a bout of an intense resistance exercise
  It will be measured through the height of the countermovement jump (CMJ)
Maximal dynamic force | 3 days (72h) after a bout of an intense resistance exercise
  It will be measured by means of a CMJ with a load
Ability to change direction | 3 days (72h) after a bout of an intense resistance exercise
  It will be measured by repeated sprint T-test

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Instituto Mixto Universitario Deporte y Salud (iMUDS), Granada
  - Facultad de Ciencias del Deporte, Granada

IPD SHARING:
Plan to Share IPD: No